CLINICAL TRIAL: NCT04119687
Title: An Open-Label, Single Ascending Dose Study to Assess the Safety and Tolerability of FX201 in Patients with Osteoarthritis of the Knee
Brief Title: Study to Evaluate the Safety and Tolerability of FX201 in Patients with Osteoarthritis of the Knee
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FX201-2019-001
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Part 1 - Open-Label, Single Ascending Dose Phase Part 2 - Open-Label, Expansion Phase to enroll additional patients in DMC-cleared dose levels by sequential assignment against a pre-defined randomized list
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose FX201 (Experimental): Single low dose FX201 injection
  Interventions: Biological: FX201
- Mid Dose FX201 (Experimental): Single mid dose FX201 injection
  Interventions: Biological: FX201
- High Dose FX201 (Experimental): Single high dose FX201 injection
  Interventions: Biological: FX201

INTERVENTIONS:
Biological: FX201 — FX201, humantakinogene hadenovec, is a novel interleukin-1 receptor antagonist (IL-1Ra) gene therapy for IA administration that is being developed for the treatment of patients with OAK.

SUMMARY:
This two-part study will be conducted in male and female patients, 30 - 80 years of age with painful OA of the index knee with Kellgren-Lawrence (K-L) Grade 2, 3 or 4.

Part 1 - Single Ascending Dose (SAD) Phase: Up to three ascending doses of FX201 will be tested in cohorts of 5-8 patients. Each patient will only receive one injection of FX201. An independent Data Monitoring Committee (DMC) will review safety and guide the conduct of the study.

Part 2 - Expansion Phase: Up to an additional 35 patients will be enrolled at each dose level reviewed by the DMC. Each patient will only receive one injection of FX201.

DETAILED DESCRIPTION:
This two-part study will be conducted in male and female patients, 30 - 80 years of age with painful OA of the index knee with Kellgren-Lawrence (K-L) Grade 2, 3 or 4.

Part 1 - SAD Phase: Up to three ascending doses of FX201 (low dose, mid dose and high dose) will be tested in cohorts of 5-8 patients. Each patient will only receive one injection of FX201. A maximum of 24 patients will be enrolled (range 15 to 24).

When a minimum of 4 weeks have elapsed since the last patient of the current cohort has been treated, all safety data will be collected and reviewed by an independent Data Monitoring Committee (DMC). After evaluating cohort safety data, the DMC will evaluate continuing the trial and initiating treatment in the next dosing cohort as well as expanding enrollment in dose level(s).

Part 2 - Expansion Phase: After the DMC has met to review safety data from each Cohort and has recommended expanding dose level(s), enrollment slots for dose levels reviewed by the DMC will be opened. A maximum of 105 patients [up to an additional 35 patients per dose level (up to 20 FX201 alone and up to 15 FX201 with IA methylprednisolone 40 mg/mL pre-treatment)].

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Male or female 30 to 80 years of age, inclusive, on the day of enrollment (Day 1)
* Body mass index (BMI) ≤ 40 kilograms per meters squared (kg/m2)
* Clinical diagnosis of OA of the knee on the American College of Rheumatology criteria (Altman, 1986) with radiologic evidence of OA (K-L Grade 2 or 3 for SAD Phase Cohort A and K-L Grade 2, 3 or 4 for SAD Phase Cohorts B and C and the Expansion Phase) at the index joint at the screening visit
* Moderate pain in the index joint
* Failed two or more types of conservative therapy for index knee osteoarthritis (e.g., structured exercise programs, topical or oral non-steroidal anti-inflammatory therapies); or failed one prior type of conservative therapy and at least one prior index knee IA treatment (corticosteroid or hyaluronic acid)
* Sexually active females and males agree to use highly effective methods of contraception

Exclusion Criteria:

* Reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease
* History of or current infection in the index knee joint
* Inability to undergo Magnetic Resonance Imaging (MRI) due to presence of surgical hardware or other foreign body in the index knee
* Unstable index knee joint (e.g., torn anterior cruciate ligament, etc.) within 12 months of Screening
* Any IA drug/biologic use within 6 months of Screening or 5 half-lives (whichever is longer) (e.g., IA corticosteroid, IA hyaluronic acid, platelet rich plasma injection, stem cells, prolotherapy and amniotic fluid injection, etc.)
* Cold or radiofrequency nerve ablation of the index knee within 12 months of Screening
* Arthroscopic or open surgery on the index knee within 12 months of Screening or planned/anticipated surgery on the index knee for the study period
* Anticipated major surgery during the study period
* Laboratory values that meet exclusion criteria
* ECG abnormality at Screening or Baseline judged clinically significant
* Use of immunomodulators, immunosuppressive, or chemotherapeutic agents within 5 years of Screening
* Use of any other investigational drug, biologic or device within 3 months of Screening
* Any systemic or local bacterial or viral infection requiring IV antibiotics or antivirals within 4 weeks of Screening or oral antibiotics or antivirals within 2 weeks of Screening
* Known allergy or sensitivity to methylprednisolone
* Any other clinically significant acute or chronic medical conditions (e.g., bleeding disorder) that, in the judgment of the Investigator, would preclude the use of an IA injection or that could compromise patient safety, limit the patient's ability to complete the study, and/or compromise the objectives of the study

Note: Other protocol defined inclusion/exclusion criteria apply.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: Incidence of treatment emergent adverse events after a single intra-articular (IA) injection of FX201 (safety and tolerability) | Baseline to Week 104
  Incidence of treatment emergent adverse events after a single intra-articular (IA) injection of FX201

SECONDARY OUTCOMES:
Secondary Outcome Measure: Characterization of the systemic biodistribution of FX201 as seen through the percentage of patients positive for FX201 at Baseline, Day 1, Day 2, Week 1, Week 2, Week 3, and Week 4 | Baseline, Day 1, Day 2, Week 1, Week 2, Week 3, Week 4
  The percentage of patients positive for FX201 at select timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Barese, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (6):
- United States (6):
  - Arizona Research Center, Phoenix, Arizona
  - Gulfcoast Research Institute, LLC, Sarasota, Florida
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - University Orthopedics Center, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta S, He T, Bajpayee AG. Recent advances in targeted drug delivery for treatment of osteoarthritis. Curr Opin Rheumatol. 2021 Jan;33(1):94-109. doi: 10.1097/BOR.0000000000000761. PMID 33229973